CLINICAL TRIAL: NCT06921642
Title: "Performance of a Simplified Inferior Vena Cava Collapsibility Methodology to Predict Preload Responsiveness (PR) in Spontaneously Breathing and Critically Ill Patients"
Brief Title: Simplified Inferior Vena Cava Collapsiblity
Acronym: CVCISIMPLIFIEE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0324
Record Dates: First submitted 2025-03-07; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Circulatory Failure
Keywords: Fluid therapy; preload responsiveness; spontaneously breathing; critically ill patient; standardized inspiratory maneuver
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Spontaneous breathing patient responding to the inclusion criteria: During a transthoracic echocardiography, the doctor will realize
  * loops on inferior vena cava in different breathing conditions :
    * non standardized spontaneous breathing
    * simplified standardized spontaneous breathing using a TRIFLOW III spirometer device. Standardized inspiration is defined by the complete ascension of the first of the three device ball.
    * deep spontaneous inspiration defined by profound inspiration during < 3 seconds without calibration of inspiratory strengh
  * measure of subaortic velocity time integral (Vti) during a passive leg raising.
  Inferior vena cava collapsibility index will be calculated using inferior vena cava diameter, at 4 cm from right atrium abutment, using the following equation: (Diameter max - diameter min)/ diameter max.
  PR will be defined by 10% increase of Vti during passive leg raising.
  Interventions: Device: Echocardiography images

INTERVENTIONS:
Device: Echocardiography images — Addition of a recording loop during routine ultrasound, during which the patient is in simplified standardized ventilation

SUMMARY:
Fluid administration is a cornerstone therapy in critically ill patient. Fluid restriction or overload can therefore change patient's outcome and mortality. Close monitoring of PR (capacity of increase the cardiac output after fluid therapy) is recommended by experts' guidelines. Few bedside simple tests are available to predict PR in spontaneously breathing patients.

A team of investigators from Lille (Roger Salengro hospital) have already showed that inferior vena cava collapsibility (cVCI) accuracy of prediction of PR is excellent in standardized sponteanous breathing patient. However, the standardized inspiration maneuver remains challenging because requiring specific and non-widely available equipment.

DETAILED DESCRIPTION:
The primary objective of this study is to confirmed the excellent accuracy of cVCI to predict PR when standardized inspiratory maneuver is simplified.

The secondary objective is to test cVCIs in different period of cardiac cycle guided by electrocardiogram.

After receiving a loyal information patients will give their non-objection. During systematic echocardiography, patients will have to breathe in different conditions in order to homogenize their inspiratory effort. This maneuver will be repeated three times.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring an evaluation of PR by echocardiography for
* Presence of at least one clinical sign of acute circulatory failure (Mean Arterial Pressure < 65 mmHg, mottling, tachycardia with Heart Rate > 90 bpm, capillary refill time > 3 sec, oliguria (urine output < 0,5 mL/kg/h over 1 hour or more))
* Noradrenaline administration
* Age > 18 years old
* Spontaneous breathing patient requiring oxygen administration without mechanical assistance

Exclusion Criteria:

* Intolerance of inspiratory maneuver defined by:

  * Clinical sign of acute respiratory failure
  * Active abdominal expiration
* Hemodynamic response of passive leg raising not evaluable:

  * Intracranial hypertension
  * Impaired transthoracic or abdominal echogenicity
  * High grade aortic insufficiency
  * Pregnancy
  * Abdominal compartment syndrome
  * Lower limb amputation
* Urgent hemodynamic therapy within half an hour
* Modification of hemodynamic support (fluid therapy or modification of catecholamine dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient hospitalized in an intensive care unit of the Medecine intensive center of Lille who respond to the inclusion criteria may be included in this trial
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Performance of simplified inferior vena cava collapsibility index to predict preload responsiveness | The echocardiographic loops used to measure cVCI and preload responsiveness will be performed on the day of inclusion refered as baseline. Precise measurements will be conducted offline within the 6 months after the end of the inclusions.
  the area under the ROC curve of the parameter of simplification of inspiratory effort in relation to the positive hemodynamic response positive haemodynamic response (cardiac preload-dependence) to a passive leg raising manoeuvre

SECONDARY OUTCOMES:
Performance of inferior vena cava collapsibility index during a deep breath (without monitoring of inspiratory strength) to predict preload responsiveness | The echocardiographic loops used to measure cVCI and preload responsiveness will be performed on the day of inclusion refered as baseline. Precise measurements will be conducted offline within the 6 months after the end of the inclusions.
  comparison of the areas under the ROC curve for the parameter simplifying inspiratory effort during tele-diastole or tele-cardiac systole
Performance of simplified inferior vena cava collapsibility index to predict preload responsiveness during different time of cardiac cycle | The echocardiographic loops used to measure cVCI and preload responsiveness will be performed on the day of inclusion refered as baseline. Precise measurements will be conducted offline within the 6 months after the end of the inclusions.
  the area under the ROC curve of the parameter of simplification of inspiratory effort in relation to the positive hemodynamic response positive haemodynamic response (cardiac preload-dependence) to a passive leg raising manoeuvre

CONTACTS AND LOCATIONS:
Locations (1):
- Lille University Hospital, Lille, France